CLINICAL TRIAL: NCT00207012
Title: Continuous Dosing Phase I Study of BMS-599626 in Patients With HER2-Expressing Advanced Solid Malignancies
Brief Title: MAD Refractory: Solid Tumor QD w/o Break
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA181-003
Record Dates: First submitted 2005-09-12; First posted 2005-09-21 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2009-01

CONDITIONS: HER2 or EGFR Expressing Advanced Solid Malignancies
MeSH Terms: interventions — (4-((1-(3-fluorophenyl)methyl)-1H-indazol-5-ylamino)-5-methylpyrrolo(2,1-f)(1,2,4)triazin-6-yl)carbamic acid 3-morpholinylmethyl ester

INTERVENTIONS:
Drug: BMS-599626

SUMMARY:
This is a continuous dosing Phase I Study of BMS-599626 in patients with HER2-expressing advanced solid malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Available for periodic follow-up
* Life expectancy of at least 3 months
* ECOG performance status score 0-1
* Histologic or cytologic diagnosis of a primary malignancy of breast, ovarian, bladder, gastric, non small cell lung or colon origin
* Tumor paraffin tissue block or 20-30 unstained slides from tumor issue block must be provided for biomarker and predictive marker analyses
* Immuno-histochemistry (IHC) analysis of tumor biopsy demonstrating 1+, 2+ or 3+ HER3 expression or EGFR expression. For patients with breast cancer tumors must be HER2 FISH positive (fluorescence in situ hybridization). This analysis may be performed by hospital laboratory
* Evidence (radiographic or tissue confirmation) that the disease is metastatic (locally advanced disease is allowable only if no surgical or local therapeutic option exists)
* Disease which has progressed on or following currently available standard therapies or for which no standard therapy exists. (Prior adjuvant or neoadjuvant therapy is permitted. Prior investigational agents are permitted)
* Measurable or non-measurable disease
* Adequate bone marrow function defined as:
* absolute neutrophil count (neutrophil and bands)
* >=1,500 cells/mm3
* platelet count >=1000,000 cells/mm3
* hemoglobin >= 9.0 g/dl
* Adequate hepatic function defined as:
* total bilirubin <= 1.5 times the institutional upper limits of normal
* alanine aminotransferase (ALT) and aspartate aminotransferase (AST)<=2.5 times the institutional upper limit of normal
* Adequate renal function defined as:
* serum creatine <=1.5 times the institutional upper normal limit
* PT-INR/PTT ,=1.5 x upper limit of normal. Prophylactic coumadin is allowed
* Serum potassium, calcium and magnesium levels within institutional normal limits
* Prior anticancer chemo-, radio-, hormonal or immunotherapy are allowed. Patients must have recovered from toxicity due to prior therapy (i.e., toxicity has resolved to baseline or is deemed irreversible). At least 4 weeks must hav elapsed since the last chemotherapy (6 weeks for nitrosoureas, mitomycin-C, and liposomal doxorubicin), immunotherapy or radiotherapy and beginning of protocol therapy. At least 2 weeks must have elapsed since last anticancer hormonal therapy or "targeted" kinase inhibitor (e.g. Herceptin)
* Men and women, ages 18 and above
* Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for at least 3 months after the study in such a manner that the risk of pregnancy is minimized
* WOCBP include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation or bilateral oophorectomy) or is not postmenopausal Even women who are using oral, implanted or injectable contraceptive hormones or mechanical products such as an intrauterine device or barrier methods (diaphragm, condoms, spermicides) to prevent pregnancy or practicing abstinence or where partner is sterile (e.g. vasectomy) should be considered to be of child bearing potential.
* WOCP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 72 hours prior to the start of study medication.

Exclusion Criteria:

* WOCBP who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for at least 3 months after the study
* WOCBP using a prohibited contraceptive method
* Women who are pregnant or breastfeeding
* Women with a positive pregnancy test on enrollment or prior to study drug administration
* Men who are unwilling or unable to use an acceptable method of birth control if their sexual partners are WOCBP for the entire study period and for at least 3 months after completion of the study
* Patients with known brain metastasis. Patients with controlled brain metastasis (no progression for 60 days following defined treatment and no neurologic signs or symptoms) will be allowed. Patients with signs or symptoms or suggestive of brain metastasis are not eligible unless brain metastasis are ruled out by CT or MRI
* A serious uncontrolled medical disorder or active infection which would impair the ability of the patient to receive protocol therapy
* Uncontrolled or significant cardiovascular disease, including:
* A myocardial infarction within 12 months
* Uncontrolled angina within 6 months
* Congestive heart failure within 4 months or left ventricular ejection fraction (LVEF) below lower limit of normal or below 45%
* Diagnosed or suspected congenital long QT syndrome
* Any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or torsade de pointes). Any patient with a history of any arrhythmia should be discussed with the bMS Medical Monitor prior to entry into the study
* Prolonged QTc interval on pre-entry electrocardiogram (>450 msec)
* Any history of second or third degree heart block (may be eligible if currently have a pacemaker)
* Heart rate <50/minute on pre-entry electrocardiogram
* Uncontrolled hypertension
* Dementia or altered mental status that would prohibit the understanding or rendering of informed consent
* Known allergy to BMS-599626 or related compound
* Investigational agents during or within 4 weeks prior to the start of protocol therapy
* Recent anticancer therapy
* Drugs (or medical condition) that are generally accepted to have a risk of causing Torsade de Pointes. Patients who have discontinued any of these medications must have a wash-out period of at least 5 days or at least 5 half-lives of the drug (whichever is greater) prior to the first dose of BMS-599626
* Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (e.g., infectious disease) illness must not be enrolled into this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45
Dates: Start 2004-05; Primary Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Determine the maximum tolerated, biologically active doses and recommended phase 2 dose(s) of BMS-599-626 when administered as a daily uninterrupted oral dose

SECONDARY OUTCOMES:
Efficacy (Best Clinical Response)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (2):
- Local Institution, Villejuif, France
- Local Institution, Barcelona, Spain